CLINICAL TRIAL: NCT04154020
Title: Treatment of Ulcers Associated With Hammer, Mallet and Claw Toe Deformities in the Diabetic Patient Setting
Acronym: TODDII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Jonas Hedegaard Andersen, Orthopedic Consultant & Clinical Assistant, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TODD II
Record Dates: First submitted 2019-09-03; First posted 2019-11-06 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer; Hammer Toe; Mallet Toe; Claw Toe
Keywords: tenotomy
MeSH Terms: conditions — Diabetic Foot; Hammer Toe Syndrome

STUDY DESIGN:
Intervention Model Description: Patients who meet all inclusion and no exclusion criteria are randomly allocated to two arms in the study. The allocation is stratified by treatment center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenotomy (Experimental): Patients allocated to this arm receive tenotomy treatment of affected toes, and standard care including offloading treatment
  Interventions: Procedure: Flexor tenotomy
- standard care (No Intervention): Patient who are randomized to this arm receive standard care including offloading treatment

INTERVENTIONS:
Procedure: Flexor tenotomy — Tenotomy(cutting) of flexor tendons is performed with needle
  Arms: Tenotomy

SUMMARY:
1. Aim Patients with diabetes, hammer, mallet and claw toes and ulcers associated with the named deformities will be randomized to tenotomy (cutting) of flexor tendons to the afflicted toes, done by needle and standard offloading or offloading alone. The effects of the surgery on time to healing of ulcers associated with the named deformities, recurrence of the ulcers, and rate of complications associated with the surgery. In addition to this all patients gait and balance will be examined before start of the study, and after 3 months, to se if there is an effect of the surgery on patients gait and balance.
2. Method A prospective randomized clinical study, which means a study were patients will be allocated randomly to surgery and standard care or standard care alone.

Patients will attend a total of up to 14 visits over a 12-month period.

3.

DETAILED DESCRIPTION:
1. STUDY RATIONAL Diabetes is one of the largest medical challenges facing the world today. 12% of the world's health budget is spent on diabetes, which is USD 673 billion (Euros 585 billion). It is estimated that a lower limb is amputated due to diabetes every 30 sec. on a global scale, and its known that 85% of all amputations are performed due to a diabetic ulcer1. In Denmark 320.000 citizens has a diabetes diagnosis, an additional 200.000 are estimated to have diabetes unknowingly, and 750.000 to have the pre-stages of diabetes2. These numbers have doubled in the past ten years and are estimated to cost DKK 86 million a day (or Euros 11.6 million a day)1. One of the complications to diabetes is the "diabetic foot syndrome", which is a result of neurological abnormalities, vascular complications or a combination of the two. Knowledge about the causes of the disease has been gathered since the late nineteenth century3. In recent years, preventive therapy has been the focus of treatment, resulting in several national and international guidelines4,5,6. Focus has been on education in self-care and awareness of risk factors, combined with "Foot-at-Risk" evaluation7, at least once a year and off-loading therapy crafted and applied by specialized personnel3,4.

   Steno Diabetes Center Copenhagen, University of Copenhagen, Denmark is a highly-specialized treatment facility focusing on the patient with diabetes. In spite of optimized treatment for patients with diabetes, and the fact that incidence of first-time ulcers in patients with type 1 and 2 diabetes is declining, the incidence of first time ulcers is still 2.6 and 8.7 per. 1000 patient years for type 1 and 2, respectively8. Diabetic foot ulcers have a known association with increased mortality, morbidity and economic burden9,10,11, at the same time most amputations in patients with diabetes are preceded by an ulcer12.

   Hammer, mallet and claw-toe deformities are some of the most common deformities associated with the diabetic foot syndrome. Prevalence has been reported between 32% and 46%13,14. These deformities are predictors of diabetic foot ulcers15,16. There are several theories on the etiology of hammer, mallet and claw toe deformities - the three classic deformities of the toes. In the diabetic patient setting, the classical theory is based on neuropathy (nerve damage associated with diabetes and other diseases), resulting in intrinsic muscle (muscles of the foot) dysfunction, changes that lead to imbalance between the flexor and extensor tendons, which in turn leads to hyperextension of the metatarsophalangeal (MTP) joint and/or flexion in the interphalangeal joints (IP), leading to the three classic deformities of the toes. The neuropathic theory is not sufficient to explain the full 4 scope of the problem, and other theories have been proposed17. In the non-diabetic patient, the neuropathic explanation is not viable, but the explanations still center on an imbalance between in- and extrinsic musculature, resulting from deformities in the foot either as flexor-substitution or stabilization deformities18. The deformities change the pressure on the plantar aspect of the foot19. These changes in pressure make specific contact point's predilection sites for ulcers. The sites have been described as tip of the toe ulcers, cock-up ulcers, kissing ulcers and plantar metatarsal ulcers20, these sites will be referred to as ulcers associated with hammer, mallet and claw toe deformities, and are defined as cock-up ulcers that are placed at the dorsal side of proximal phalangeal joint of toes 2-5 and inter phalangeal joint of the hallux. A tip of the toe ulcer is placed at the pulpa of the affected toe. Metatarsal ulcers are placed at the plantar aspect of the distal head of the metatarsal bone of the involved toe. Kissing ulcers, which are placed between toes, and is due to pressure from the deformed toe/toes.

   The treatment of hammer, mallet and claw toe deformities in diabetes has classically consisted of offloading in the form of shoes, insoles and/or orthosis (i.e. silicone spacers, felt pads etc.) or flexor tendon tenotomy (cutting tendons) done by scalpel. Several studies on flexor tenotomies performed with scalpel have been performed21,22; all have reported acceptable or positive results on ulcer healing and low complication rates, including one study from our own institute23. At Diabetic Foot Study Group 2018 we presented unpublished results from a study showing that tenotomy done by needle has comparable results to the classical scalpel. However, no study has, to our knowledge, been published comparing conservative treatment with surgical approach to these deformities, let alone randomized controlled trials (RCT). At the same time no studies have, to our knowledge, looked at the effect on plantar pressure (pressure profile of the foot) and balance post flexor tenotomy in the above-mentioned setting.
2. WHAT DOES THIS TRIAL ADD TO CURRENT KNOWLEDGE? This is to our knowledge the first RCT looking at flexor tenotomies compared to conservative treatment. At the same time this is the first study looking at needle flexor tenotomies, as opposed to the classic tenotomies done by scalpel. The effect of flexor tenotomy on the balance of patients with diabetes has not been described earlier.
3. HYPOTHESIS We hypothesize that treating ulcers associated with hammer, mallet and claw toe deformities in patients with type 1 and 2 diabetes with needle tenotomy is a safe and effective treatment, and superior to offloading (conservative) treatment done by silicon spacer, insoles, felt, and/or therapeutic sandals.

   I addition we hypothesize that needle tenotomy performed as a treatment for ulcers associated with hammer, mallet and claw toe deformities in patients with type 1 and 2 diabetes will not affect the patients balance or gait significantly.
4. AIM This study is a randomized controlled trial (RCT) . The aim of the RCT is to evaluate the effect of needle tenotomy when treating hammer, mallet and claw toe deformities and an associated ulcer in patients with diabetes.
5. Study 5.1 Design A prospective RCT involving patients with diabetes as well as one of the three deformities and an active ulcer associated with the mentioned deformities.

   5.2 Patients Note Patients who don't meet the additional inclusion and exclusion criteria for gait and balance will be excluded from gait and balance but not the rest of the study. Conversely patients who don't meet inclusion and exclusion criteria other than those additional for gait and balance will not be eligible for enrollment in any part of the study.

   Discontinuation of patients
   * Patient discontinues assigned treatment for any reason, while not fulfilling one of the studies accepted endpoints
   * Patient incurs a serious adverse event (SAE), defined as death or sepsis related to the study procedure
   * Investigator decides to discontinue patient due to health or compliance reasons
   * Patient misses 3 consecutive visits
   * Patient misses 5 or more visits during the full treatment period Patients who discontinue the study early will be invited to have a clinical visit before being discontinued.

   Patients that are discontinued will revert to their normal treatment plan, and continue in their respective clinics.

   5.3 Statistical Analysis Plan

   Sample-size The calculation is based on a Type 1 error rate of 5%, and a power of 80%. The primary endpoint is time-to-heal of ulcer associated with hammer, mallet or claw toe deformity. The mean of the intervention group is set at 4 weeks, which is the average time to healing we observed in a pilot study done on needle tenotomies at our institute24, while the mean of the control group is set at 10 weeks, which has been reported by Zimny when evaluating diabetic foot ulcers treated with standard care25,26. However, time-to-heal, when looking at the diabetic foot ulcer, is dependent on multiple factors like size, etiology and patient co-morbidities, therefore the standard deviation is set at 10. The clinical minimal relevant difference (miredif) for time-to-heal is set at 6 weeks. 6 weeks shorter time-to-heal, is seen as clinically relevant difference, on based on clinical experience, and a goal of time to heal at 4 weeks compared to the above reported 10 week average healing time attained with standard care31,32.

   The calculator used is a 2 means, 2 sample, 2-sided equality calculator. With the above described parameters, the sample size is 44 patients, which due to an expected dropout of 10% will be extended to 50 patients.
6. PERSPECTIVE

   The results of these studies will allow us to evaluate if there is a clinical advantage in performing tenotomies. Several studies have shown that tenotomies done by scalpel are safe and that most ulcers heal27,28, but none have compared tenotomies with standard care. Our hypothesis is that patients with ulcers associated with hammer, mallet and claw toe deformities will heal faster when treated by tenotomy. At the same time, unpublished data from our institute show that tenotomy done by needle has comparable results to tenotomy done by scalpel. If this minimal invasive procedure, that can easily be performed in an everyday clinical setting, can lead to significant reductions in healing times, there is a potential for significant reductions in socioeconomic costs.
7. QUALITY CONTROL AND MONITORING

   The studies will be performed in accordance with the Helsinki Declaration, International Council for Harmonization of technical requirements for pharmaceuticals for human use (ICH) Guidelines for good Clinical Practice (GCP)29 and after approval by the The National Committee on Health Research Ethics and the Data Monitoring Board in Denmark. The study will be registered on http://www.clinicaltrials.gov/.

   Permission for a third person to have access to patient data will be obtained at screening visit. Investigators will provide access to source data and relevant documents in connection with monitoring, inspections, and audits to all relevant authorities.
8. ETHICAL CONSIDERATIONS AND DATA SAFETY

   8.1 Ethics The study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki 1996 and the principles of GCP30 8.1 Ethical committee approval The appropriate approval from a local Danish ethical committee will be obtained before start of trial, and their guidelines will be followed throughout the process. Patients will receive oral and written information on the study, before being required to sign an informed consent paper.

   8.2 Personal data usage and protection The appropriate approval from the Danish data protection agency will be obtained before the study commences, and their guidelines will be followed throughout the process. All patient data will be stored and treated in accordance with regulation 2016/679 from the European parliament on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, dated 27 April 201631, and the Danish amendment to regulation 2016/67932.

   8.3 Patient Perspective and Conclusion Patients enrolled in this study will receive a treatment that is already implemented in our and several other clinics, and the unpublished data from our retrospective study and the formerly published data on tenotomies, points towards tenotomies being a safe and effective treatment of hammer, mallet and claw toes, with a low risk of complications for patients with diabetes. The enrolled patients will in addition receive a gait and balance analysis that can be used as a diagnostic tool to help in treatment generally. Patients who don't receive intervention in the form of tenotomies in the study, will receive standard offloading and ulcer treatment, and be offered to undergo tenotomy after completing 10 weeks observation in the study if relevant in addition they will be offered a gait and balance examination with mentioned benefits. In conclusion the patients enrolled in the study will receive a treatment with potential benefits for them, and a low risk of complications making the study ethically sound.
9. DISSEMINATION OF RESULTS The study is initiated by Peter Rossing. Data is owned by the investigators. Positive, inconclusive as well as negative study results will be published in both national and international oral and written presentations as well as peer-reviewed international scientific journals. If data against expectations are not published in international journals, positive as well as negative study results will be published on a public website, for example www.clinicaltrials.gov.
10. PATIENT INFORMATION

10.1 Written Information All patients will receive information detailing the project, written information on their rights as Participants in research projects from the Danish ethics committee33, and written information on the procedure, potential unintended side effects, and what to expect after the operation.

10.2 Verbal Information All patients will be informed in layman's terms on the details of the operations, potential unintended side effects, and what to expect after the operation.

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18 years or above
* Type 1 or 2 diabetes
* Hammer, mallet or claw toe deformity as judged by investigator
* Ulcer associated with above mentioned deformities
* Able to understand written and oral information
* Ability to follow planned visits and treatment
* Able to provide informed consent in Danish and/or English

Exclusion Criteria

* Revascularization procedure in the affected limb planned, or undertaken within the 4 weeks prior to screening
* Hammer, claw and mallet toe that are completely rigid in both MTP and IP joints
* Toe blood pressure lower than 30mmHg
* Infections of the foot ulcer needing surgical treatment
* Prior major amputations on affected or ipsilateral leg
* Other corrective operation is indicated to treat patients foot deformities as deemed by investigator
* Current treatment with cytotoxic drugs or with systemically administered glucocorticoids
* Treatment of foot ulcers with growth factors, stem cells or equivalent preparations within the 8 weeks prior to screening
* Likely inability to comply with the need for planned visits because of planned activity
* Participation in another interventional clinical foot ulcer-healing trial within the 4 weeks prior to screening
* Prior enrolment in this trial
* Judgement by the investigator that the patient does not have the capacity to understand the study procedures or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Mean time to healing of ulcers(s) in treated limb | Measured at visits (1,3, 5, 7, 9, 10 weeks and 3, 6 and 12 months)
  Measured in days

SECONDARY OUTCOMES:
Mean time to healing of incision sites | Measured at visits (1,3, 5, 7, 9, 10 weeks and 3, 6 and 12 months)
  Measured in days
Incidence of minor amputations | 1 year
  Incidence of minor amputations
Incidence of major amputations | 1 year
  Incidence of major amputations
Plantar pressure profile | 3 months
  Measured in mmhg from the gait analysis
trembling | 3 months
  mean COP velocity
Rambling | 3 months
  measured in COP range and sway path length
incidence of secondary infection | 1 year
  Incidence of infection during observation period, as demmed by investigator
Pain in treated limb, associated with tenotomy | 1 year
  Patient reported pain associated with treatment
Transfer lesion incidence | 1 year
  Transfer lesions defined as impending ulcers or actual ulcers at anatomical sites associated with hammer, mallet and claw toes in patients with diabetes, on non-treated hammer, mallet and claw toes after surgical treatment),
Recurrence of ulcers on the treated limb | 1 year
  Measured in incidence of recurrent ulcers, defined as ulcer in same anatomical position as treated ulcer after complete healing
Incidence of new ulcers on feet | 1 year
  Measured in incidence of new ulcers, defined as ulcer in different anatomical position than the treated ulcer(s) and associated with hammer, mallet or claw toes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Prof MD, Study Director — Steno Diabetes Cneter Copenhagen
Locations (3):
- Denmark (3):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Hospitalerne i Nordsjælland Hillerød Hospital Ortopædkirurgisk afdeling, Hillerød
  - Videncenter for Sårheling Bispebjerg Hospital, København NV

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT04154020/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04154020/ICF_000.pdf